CLINICAL TRIAL: NCT05191732
Title: The Therapeutic Effect of Autologous Platelet-Rich Plasma Versus Bone Marrow Concentrate in Anterior Cruciate Ligament Reconstruction - A Prospective, Double-Blind Randomized Controlled Study
Brief Title: Effect of PRP Versus BMC in Anterior Cruciate Ligament Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Collaborators: Ministry of Health and Welfare, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KMUHIRB-F(I)-20170122
Record Dates: First submitted 2021-09-30; First posted 2022-01-13 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2021-09

CONDITIONS: Anterior Cruciate Ligament Reconstruction
Keywords: Anterior cruciate ligament reconstruction; Platelet-Rich Plasma; Bone marrow concentrate; Hamstring tendon

STUDY DESIGN:
Intervention Model Description: To investigate the result of clinical functional scoring, MRI, and biomechanical study between PRP augmentation, PRP+BMC augmentation and traditional ACL reconstruction.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PRP augmentation ACL reconstruction group (Experimental): Platelet-rich plasma (PRP) (Dosage form: APA-15)
  Interventions: Combination Product: Platelet-Rich Plasma; Bone marrow concentrate
- PRP+BMC augmentation ACL reconstruction group (Experimental): Bone marrow concentrate (BMC) (Dosage form: APA-15Q)
  Interventions: Combination Product: Platelet-Rich Plasma; Bone marrow concentrate
- Traditional ACL reconstruction group (No Intervention): No intervention

INTERVENTIONS:
Combination Product: Platelet-Rich Plasma; Bone marrow concentrate — Platelet-rich plasma (PRP) (Dosage form: APA-15) Bone marrow concentrate (BMC) (Dosage form: APA-15Q)
  Arms: PRP augmentation ACL reconstruction group; PRP+BMC augmentation ACL reconstruction group

SUMMARY:
Anterior cruciate ligament (ACL) is an important stabilizer of knee during daily activity and exercise. The ruptured ACL need to be reconstructed by a new tendon graft which passed the bone tunnel and joint during operation. How to enhance the tendon graft to bone tunnel healing is critical important to prevent recurrent ligament laxity, avoid secondary osteoarthritis, and achieve early return to sports and work.

Platelet Rich Plasma (PRP)，harvest from peripheral blood, is rich in multiple growth factors(i.e. VEGF, PDGD, TGFB, IGF, EGF) which help the injured tissue regeneration. Bone marrow stem cell has been demonstrated to enhance the injured tissue repair both in vitro and in vivo study.

However, there is no prospective study in comparing the PRP and BMC to enhance interfacial healing between graft and bone tunnel in ACL reconstruction. Investigators hypothesize that the combination of PRP and BMC has synergetic effect in interfacial healing in ACL reconstruction.

Aim of this study： To investigate the result of clinical functional scoring, MRI, and biomechanical study between PRP augmentation, PRP+BMC augmentation and traditional ACL reconstruction.

DETAILED DESCRIPTION:
Anterior cruciate ligament (ACL) is an important stabilizer of knee during daily activity and exercise. According to literature, there are 100,000- 200,000 ACL tear case annually in US. The patients with ACL tear will sustain with joint pain, muscle weakness, giving way sensation, other knee ligaments or meniscus injury, and consequent osteoarthritis change. However, the ruptured ACL cannot heal by itself due to limited vascularity supply, intraarticular inflammatory factors which inhibit the ACL cells migration and proliferation. The ruptured ACL need to be reconstructed by a new tendon graft which passed the bone tunnel and joint during operation. How to enhance the tendon graft to bone tunnel healing is critical important to prevent recurrent ligament laxity, avoid secondary osteoarthritis, and achieve early return to sports and work.

Platelet Rich Plasma (PRP)，harvest from peripheral blood, is rich in multiple growth factors(i.e. VEGF, PDGD, TGFB, IGF, EGF) which help the injured tissue regeneration. The PRP has been applied in treating tendinitis, osteoarthritis, cartilage injury, and bone nonunion. Bone marrow contains lots of stem cell and progenitor cells with capability of self-renewal and multi-differentiation. Bone marrow stem cell has been demonstrated to enhance the injured tissue repair both in vitro and in vivo study. The bone marrow concentrate (BMC) can be isolated from the bone marrow through the centrifuge procedure at one time which contains multiple stem cells. The bone marrow can regenerate itself around 1 week.

In recent years, many authors uses the combination of RPP and BMC to treat injured tissue. However, there is no prospective study in comparing the PRP and BMC to enhance interfacial healing between graft and bone tunnel in ACL reconstruction. Investigators hypothesize that the combination of PRP and BMC has synergetic effect in interfacial healing in ACL reconstruction.

The purpose of this study is to investigate the clinical outcome of autologous PRP, and combined BMC+PRP in tendon graft augmentation in the ACL reconstruction surgery with functional score and MRI evaluation. Investigators will analyze the therapeutic effect using one-way ANOVA. To investigate the result of clinical functional scoring, MRI, and biomechanical study between PRP augmentation, PRP+BMC augmentation and traditional ACL reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* Age ≧ 20 year-old
* the patient has been confirmed ACL rupture and the reconstruction is indicated
* sign IRB and operation consent

Exclusion Criteria:

* combined other ligament or extremities injury
* prior the same knee surgery
* open wound or operation history at knee joint
* Severe knee osteoarthritis
* history of multiple joint arthritis or rheumatoid arthritis
* Systemic diseases (infections, malignancies, immunodepression)
* patients with bleeding tendency, anticoagulant or antiaggregant therapies
* patients with Hb values < 11 g/dl and/or platelet values < 150,000/mm
* refuse to sign Informed Consent Form and operation consent

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-08-03 (Actual); Primary Completion 2020-07-04 (Actual); Study Completion 2020-07-04 (Actual)

PRIMARY OUTCOMES:
X-ray | preoperative
  X-ray to evaluate the joint space, graft to bone healing status and graft incorporation.
X-ray | 3 months after ACL reconstruction.
  X-ray to evaluate the joint space, graft to bone healing status and graft incorporation.
X-ray | 6 months after ACL reconstruction.
  X-ray to evaluate the joint space, graft to bone healing status and graft incorporation.
X-ray | 12 months after ACL reconstruction.
  X-ray to evaluate the joint space, graft to bone healing status and graft incorporation.
MRI | preoperative
  MRI to evaluate the joint space, graft to bone healing status and graft incorporation.
MRI of operated knee | 3 months after ACL reconstruction.
  MRI to evaluate the joint space, graft to bone healing status and graft incorporation.
MRI of operated knee | 6 months after ACL reconstruction.
  MRI to evaluate the joint space, graft to bone healing status and graft incorporation.
MRI of operated knee | 12 months after ACL reconstruction.
  MRI to evaluate the joint space, graft to bone healing status and graft incorporation.
Lysholm score | preoperative
  Lysholm score to evaluate the knee function recovery
Lysholm score | 3 months after ACL reconstruction.
  Lysholm score to evaluate the knee function recovery
Lysholm score | 6 months after ACL reconstruction.
  Lysholm score to evaluate the knee function recovery
Lysholm score | 12 months after ACL reconstruction.
  Lysholm score to evaluate the knee function recovery
IKDC 2000 | preoperative
  IKDC 2000 to evaluate the knee function recovery
IKDC 2000 | 3 months after ACL reconstruction.
  IKDC 2000 to evaluate the knee function recovery
IKDC 2000 | 6 months after ACL reconstruction.
  IKDC 2000 to evaluate the knee function recovery
IKDC 2000 | 12 months after ACL reconstruction.
  IKDC 2000 to evaluate the knee function recovery
Muscle power (N.m/kg) | preoperative
  muscle power test by Biodex System 3 Pro
Muscle power (N.m/kg) | 3 months after ACL reconstruction.
  muscle power test by Biodex System 3 Pro
Muscle power (N.m/kg) | 6 months after ACL reconstruction.
  muscle power test by Biodex System 3 Pro
Muscle power (N.m/kg) | 12 months after ACL reconstruction.
  muscle power test by Biodex System 3 Pro
Proprioception (degree) | preoperative
  Proprioception test by Biodex System 3 Pro
Proprioception (degree) | 3 months after ACL reconstruction.
  Proprioception test by Biodex System 3 Pro
Proprioception (degree) | 6 months after ACL reconstruction.
  Proprioception test by Biodex System 3 Pro
Proprioception (degree) | 12 months after ACL reconstruction.
  Proprioception test by Biodex System 3 Pro

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Hsi Chou, PhD, Principal Investigator — Kaohsiung Medical University Chung-Ho Memorial Hospital
Locations (1):
- Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.